CLINICAL TRIAL: NCT07020221
Title: A Phase 1/2, Open-label Study of VS-7375, a KRAS G12D (ON/OFF) Inhibitor, as Monotherapy and in Combination, in Patients With Advanced KRAS G12D-Mutated Solid Tumors
Brief Title: A Phase 1/2 Study of VS-7375 in Patients With KRAS G12D-Mutated Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-7375-101
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non Small Cell Lung Cancer; Colorectal Cancer; Solid Tumor, Adult; G12D Mutated KRAS
Keywords: KRAS G12D mutation; Solid tumors; Non Small Cell Lung Cancer; Lung Cancer; Colorectal Cancer; Metastatic Cancer; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; NSCLC; CRC; PDAC; Pancreatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; KRAS; RAS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms; Gastrointestinal Neoplasms | interventions — Cetuximab; Carboplatin; Pemetrexed; pembrolizumab; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- VS-7375 Dose Escalation (Experimental): To determine the recommended phase 2 dose (RP2D) for VS-7375 in patients with advanced solid tumors harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375
- Cetuximab + VS-7375 Dose Escalation (Experimental): To determine the recommended phase 2 dose (RP2D) for cetuximab + VS-7375 in patients with advanced solid tumors harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Cetuximab
- VS-7375 Recommended Phase 2 Dose Expansion (Experimental): To determine the efficacy of VS-7375 at the recommended phase 2 dose (RP2D) in patients with advanced PDAC, NSCLC, or solid tumors harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375
- Cetuximab + VS-7375 Recommended Phase 2 Dose Expansion (Experimental): To determine the efficacy of cetuximab +VS-7375 at the recommended phase 2 dose (RP2D) in patients with advanced CRC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Cetuximab
- VS-7375 + Carboplatin/Pemetrexed/Pembrolizumab Dose Escalation (Experimental): To determine the recommended phase 2 dose (RP2D) for VS-7375 in combination with carboplatin/pemetrexed/pembrolizumab in patients with advanced 1L NSCLC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Carboplatin + Pemetrexed + Pembrolizumab
- VS-7375 + Carboplatin/Pemetrexed/Pembrolizumab Dose Expansion (Experimental): To determine the efficacy of VS-7375 in combination with carboplatin/pemetrexed/pembrolizumab at the RP2D in patients with advanced 1L NSCLC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Carboplatin + Pemetrexed + Pembrolizumab
- VS-7375 + Gemcitabine/Nab-Paclitaxel Dose Escalation (Experimental): To determine the recommended phase 2 dose (RP2D) for VS-7375 in combination with gemcitabine/nab-paclitaxel in patients with advanced PDAC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Gemcitabine + Nab-paclitaxel
- VS-7375 + Gemcitabine/Nab-Paclitaxel Dose Expansion (Experimental): To determine the efficacy of VS-7375 in combination with gemcitabine/nab-paclitaxel at the RP2D in patients with advanced PDAC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Gemcitabine + Nab-paclitaxel
- VS-7375 + Gemcitabine Dose Escalation (Experimental): To determine the RP2D for VS-7375 in combination with gemcitabine in patients 75 years or older with advanced PDAC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Gemcitabine
- VS-7375 + Gemcitabine Dose Expansion (Experimental): The determine the efficacy of VS-7375 in combination with gemcitabine at the RP2D in patients 75 years or older with advanced PDAC harboring a KRAS G12D mutation.
  Interventions: Drug: VS-7375; Drug: Gemcitabine

INTERVENTIONS:
Drug: VS-7375 — VS-7375 is a highly selective oral, non-covalent, small molecule KRAS G12D (ON/OFF) inhibitor.
Drug: Cetuximab — Cetuximab is a monoclonal antibody targeting the epidermal growth factor receptor (EGFR).
  Other Names: Erbitux
  Arms: Cetuximab + VS-7375 Dose Escalation; Cetuximab + VS-7375 Recommended Phase 2 Dose Expansion
Drug: Carboplatin + Pemetrexed + Pembrolizumab — A combination therapy regimen used as a first-line treatment for advanced non-squamous non-small cell lung cancer.
  Arms: VS-7375 + Carboplatin/Pemetrexed/Pembrolizumab Dose Escalation; VS-7375 + Carboplatin/Pemetrexed/Pembrolizumab Dose Expansion
Drug: Gemcitabine — A chemotherapy used for the treatment of several types of cancer including advanced or metastatic pancreatic ductal adenocarcinoma.
  Arms: VS-7375 + Gemcitabine Dose Escalation; VS-7375 + Gemcitabine Dose Expansion
Drug: Gemcitabine + Nab-paclitaxel — A chemotherapy regimen used for the treatment of advanced or metastatic pancreatic ductal adenocarcinoma.
  Arms: VS-7375 + Gemcitabine/Nab-Paclitaxel Dose Escalation; VS-7375 + Gemcitabine/Nab-Paclitaxel Dose Expansion

SUMMARY:
This study will assess the safety and efficacy of VS-7375 alone and in combination in patients with advanced solid tumors harboring a KRAS G12D-mutation.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals ≥18 years of age.
* Agreement to sign and date an informed consent form (ICF) approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Histologic or cytologic evidence of locally advanced unresectable or metastatic solid tumor harboring a KRAS G12D mutation.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ function
* Adequate cardiac function
* Recovered from all AEs due to previous therapies to Grade ≤1 or baseline.
* Agreement to use highly effective contraception

Key Exclusion Criteria:

* Underwent major surgical procedure as defined by the Investigator, other than for diagnosis, within 4 weeks prior to Cycle 1 Day 1,
* Receipt of chemotherapy, targeted therapy, or radiotherapy (excluding palliative radiation) within 4 weeks or 5 half-lives, whichever is shorter, or immunotherapy within 4 weeks prior to Cycle 1 Day 1
* Treatment with any investigational drug at least 4 weeks or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1.
* History of treatment with direct and specific KRAS G12D inhibitors.
* Symptomatic, untreated, or actively progressing known central nervous system (CNS) metastases.
* Inability to swallow oral medications.
* Evidence or history of uncontrolled, clinically significant hematological, renal, hepatic, endocrine, pulmonary, gastrointestinal, cardiovascular, psychiatric, coagulation, neurologic, dermatologic, autoimmune, or allergic disease
* Individuals who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Part A: To characterize the safety, tolerability, and AE profile of escalating doses of VS-7375 | Up to 2.5 years
  To characterize the safety, tolerability, and AE profile of escalating doses of VS-7375 administered on a daily oral schedule in participants with advanced solid tumors harboring a KRAS G12D mutation.
  Proportion/number of participants with AEs, TEAEs, TRAEs, SAEs, DLTs, and dose interruptions/reductions.
Part A: To identify the MTD or MFD | Cycle 1 (each cycle is 21 days)
  To identify the MTD or MFD using a BOIN design and recommend a dose for subsequent studies of VS-7375 on a daily oral schedule in participants with any KRAS G12D-mutated solid tumor.
  Proportion/number of participants with DLTs during the DLT assessment period (through C1D21).
Part B: To evaluate the preliminary anticancer activity of the optimal VS-7375 regimen | Up to 2.5 years
  To evaluate the preliminary anticancer activity of the optimal VS-7375 regimen identified from Part A in participants with advanced KRAS G12D-mutated PDAC (cohort B1), NSCLC (cohort B2), and other solid tumors (cohort B3).
  Confirmed ORR, PFS rate, unconfirmed PR and CR rates, DCR, DOR, and PFS per RECIST v1.1.
  Overall Survival
Part C: To characterize the safety, tolerability, and AE profile of VS-7375 in combination regimens. | From enrollment to the end of treatment; an average of 9 months
  To characterize the safety, tolerability, and AE profile of VS-7375 in the following combination regimens in participants with any solid tumor harboring a KRAS G12D mutation.
  * 2L+ therapy in combination with cetuximab in participants with any advanced or metastatic solid tumor harboring a KRAS G12D mutation
  * 1L therapy in combination with carboplatin, pembrolizumab, and pemetrexed in participants with previously untreated metastatic NSCLC
  * 2L+ therapy in combination with gemcitabine and nab-paclitaxel in participants with metastatic PDAC
  * 1L therapy in combination with gemcitabine in participants aged 75 years or older with previously untreated metastatic PDAC.
  Proportion/number of participants with AEs, TEAEs, TRAEs, SAEs, DLTs, and dose interruptions/reductions.
Part C: To identify a recommended dose for subsequent studies of combination dosed VS-7375. | Cycle 1 (each cycle is 21 or 28 days)
  To identify a recommended dose for subsequent studies of combination dosed VS-7375.
  Proportion/number of participants with DLTs during the DLT assessment period (through end of Cycle 1).
Part D: To determine the preliminary anticancer activity of the optimal regimen of VS-7375 as identified in Part C | Up to 2.5 years
  To determine the preliminary anticancer activity of the optimal regimen of VS-7375 as identified in Part C as:
  * 2L+ therapy in combination with cetuximab in participants with metastatic colorectal adenocarcinoma
  * 1L therapy in combination with carboplatin, pembrolizumab, and pemetrexed in participants with previously untreated metastatic NSCLC
  * 2L+ therapy in combination with gemcitabine and nab-paclitaxel in participants with metastatic PDAC
  * 1L therapy in combination with gemcitabine in participants aged 75 years or older with previously untreated metastatic PDAC.
  Confirmed ORR, PFS rate, unconfirmed PR and CR rates, DCR, DOR, and PFS per RECIST v1.1.
  Overall survival

SECONDARY OUTCOMES:
Part A: To characterize the PK of VS-7375 as 2L+ monotherapy administered on a daily oral schedule | Up to 2.5 years
  To characterize the PK of VS-7375 as 2L+ monotherapy administered on a daily oral schedule in participants with any KRAS G12D-mutated solid tumor.
  Cmax derived from plasma concentrations of VS-7375.
Part A: To evaluate the preliminary anticancer activity of VS-73753 as 2L+ monotherapy | Up to 2.5 years
  To evaluate the preliminary anticancer activity of VS-7375 as 2L+ monotherapy in participants with any KRAS G12D-mutated solid tumor.
  Confirmed ORR, unconfirmed PR and CR rates, DCR, and DOR per RECIST v1.1.
Parts B and D: To characterize the safety, tolerability, and AE profile of the recommended VS-7375 regimens from Part A and Part C | Up to 2.5 years
  To characterize the safety, tolerability, and AE profile of the recommended VS-7375 regimens from Part A (VS-7375 monotherapy) and Part C (VS-7375 in combination with other systemic therapies), administered on a daily oral schedule in participants with KRAS G12D-mutated solid tumors.
  Proportion/number of participants with AEs, TEAEs, TRAEs, SAEs, DLTs, and dose interruptions/reductions.
Parts B, C, and D: To continue to evaluate the PK of VS-7375 as monotherapy and in combination with other systemic therapies | Up to 2.5 years
  To continue to evaluate the PK of VS-7375 as monotherapy and in combination with other systemic therapies in participants with KRAS G12D-mutated advanced solid tumors.
  Cmax derived from plasma concentrations of VS-7375.
Part C: Cohort C3: To evaluate the impact of VS-7375 on nab-paclitaxel PK | Up to 2.5 years
  To evaluate the impact of VS-7375 on nab-paclitaxel PK in cohort C3.
  Change in nab-paclitaxel exposure in the presence and absence of VS-7375.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No